CLINICAL TRIAL: NCT07056556
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of BL-M09D1 for Injection in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer and Other Solid Tumors
Brief Title: A Study of BL-M09D1 in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M09D1-102
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer; Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-M09D1 (Experimental): Participants receive BL-M09D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M09D1

INTERVENTIONS:
Drug: BL-M09D1 — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is an open-label, multicenter, dose-escalation and cohort-expansion, non-randomized Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy of BL-M09D1 for injection in patients with locally advanced or metastatic non-small cell lung cancer and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age: ≥18 years and ≤75 years (Phase Ia); ≥18 years (Phase Ib);
4. Expected survival time ≥3 months;
5. Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer or other solid tumors that have failed standard treatment;
6. Willing to provide archived or fresh tumor tissue samples from primary or metastatic lesions within the past 2 years;
7. Must have at least one measurable lesion as defined by RECIST v1.1;
8. ECOG performance status score of 0 or 1;
9. Toxicities from prior anti-tumor therapy have recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction (LVEF) ≥50%;
11. Organ function levels must meet the requirements;
12. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5 × upper limit of normal (ULN);
13. Urine protein ≤2+ or ≤1000mg/24h;
14. For premenopausal women with childbearing potential, a serum pregnancy test must be negative within 7 days before starting treatment, and they must not be breastfeeding. All enrolled patients (regardless of gender) must use adequate barrier contraception throughout the treatment period and for 6 months after treatment completion;
15. The subject has the ability and willingness to comply with the visits, treatment plans, laboratory tests, and other study-related procedures specified in the protocol.

Exclusion Criteria:

1. Received chemotherapy, biological therapy, immunotherapy, etc., within 4 weeks or 5 half-lives before the first dose;
2. History of severe cardiac disease;
3. Prolonged QT interval, complete left bundle branch block, or third-degree atrioventricular block;
4. Active autoimmune or inflammatory diseases;
5. Diagnosed with another malignancy within 5 years before the first dose (except cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix);
6. Unstable thrombotic events requiring therapeutic intervention within 6 months before the first dose;
7. Poorly controlled hypertension;
8. Poorly controlled diabetes mellitus;
9. History of interstitial lung disease (ILD) requiring steroid therapy, current ILD, or ≥Grade 2 radiation pneumonitis;
10. Concurrent pulmonary diseases resulting in clinically severe respiratory impairment;
11. Active central nervous system metastases;
12. History of allergy to recombinant humanized antibodies or human-mouse chimeric antibodies, or hypersensitivity to any excipient of BL-M09D1;
13. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
14. Cumulative dose of anthracyclines >360 mg/m² in prior (neo)adjuvant anthracycline therapy;
15. Positive for human immunodeficiency virus (HIV) antibody, active tuberculosis, active hepatitis B virus (HBV) infection, or active hepatitis C virus (HCV) infection;
16. Active infections requiring systemic treatment within 4 weeks before the first study drug administration;
17. Pleural, peritoneal, pelvic, or pericardial effusion requiring drainage and/or symptomatic within 4 weeks before the first study drug administration;
18. Participation in another clinical trial within 4 weeks or 5 half-lives before the first dose;
19. Pregnant or lactating women;
20. Other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M09D1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M09D1 . The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M09D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-M09D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-M09D1 will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-M09D1 will be investigated.
AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to approximately 24 months
  CL in the serum of BL-M09D1 per unit of time will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-M09D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-M09D1 antibody (ADA) will be investigated.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib: Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China